CLINICAL TRIAL: NCT07066813
Title: T-Staging Strategies and Their Prognostic and Therapeutic Significance in Lung Cancer With Cystic Airspaces: A Retrospective Cohort Study
Brief Title: Staging Strategies and Their Association With Prognosis and Therapy in Lung Cancer With Cystic Airspaces
Status: Recruiting | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Chen Chen, Associate Professor, Second Xiangya Hospital of Central South University
Other Study IDs: LYEC2025-K0017
Record Dates: First submitted 2025-07-05; First posted 2025-07-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer Associated With Cystic Airspaces

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: radiologic T stage based on the maximum tumor diameter including cystic components
- group 2: radiologic T stage based on the diameter of the solid/invasive portion only
- group 3: pathologic T stage derived from the resected specimen

SUMMARY:
The goal of this observational study is to determine the most accurate tumor size measurement method for T-staging and prognostic assessment in lung cancer with cystic airspaces (LCCA). The main questions it aims to answer are:

* What is the optimal T-staging approach for accurately classifying lung cancer with cystic airspaces （LCCA) and predicting patient outcomes?
* How do imaging features of cystic lesions correlate with their pathological characteristics?
* What is the relationship between imaging features of cystic airspace-associated lesions and patient prognosis?
* Can optimizing the T-staging method improve clinical decision-making in patients with LCCA?

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-small cell lung cancer (NSCLC), as verified by biopsy or postoperative pathological examination;
2. Patients who have undergone surgical lung resection;
3. Patients with complete preoperative chest CT imaging data;
4. Preoperative chest CT showing a well-defined gas-containing (air-filled) cystic component within the tumor.

Exclusion Criteria:

1. History of pulmonary diseases that could produce cystic lung lesions (e.g., tuberculosis, pulmonary fungal infections, bullae, emphysema, Lymphangioleiomyomatosis [LAM], or Birt-Hogg-Dubé [BHD] syndrome);
2. Systemic anti-tumor therapies, including chemotherapy, radiotherapy, or targeted therapies (such as monoclonal antibodies, small-molecule tyrosine kinase inhibitors, among others), were administered prior to enrollment;
3. Patients with concurrent other malignancies;
4. Patients with missing or poor-quality preoperative chest CT imaging data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with LCCA who underwent surgical treatment in the Second Xiangya Hospital of Central South University
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
DFS | From enrollment to the end of surgery for 5 years
  Disease-Free Survival
OS | From enrollment to the end of surgery for 5 years
  Overall Survival

SECONDARY OUTCOMES:
Rate of T-stage reclassification | From enrollment to the end of surgery for 5 years
  T-stage reclassification
AI-based extraction of radiologic characteristics of cystic airspace-associated lesions | From enrollment to the end of surgery for 5 years
  Machine learning was employed to extract and analyze the radiologic characteristics of cystic airspace-associated lesions.
AI to extract and analyze pathological features | From enrollment to the end of surgery for 5 years
  Machine learning was employed to extract and analyze pathological features
Oncogenic driver genetic alterations | From enrollment to the end of surgery for 5 years
  Results of driver gene mutation testing
Receipt of postoperative adjuvant therapy | From enrollment to the end of surgery for 5 years
  Postoperative adjuvant therapy was ascertained from medical records

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No